CLINICAL TRIAL: NCT05374213
Title: Effects of a Virtual Mindfulness-based Intervention for Depression and Anxiety in a Community Psychiatric Sample
Brief Title: Virtual Mindfulness Intervention RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Joseph Brant Hospital (Other)
Responsible Party: Principal Investigator, Dr. Neil Rector, Senior Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3181
Record Dates: First submitted 2021-07-15; First posted 2022-05-16 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2022-05

CONDITIONS: Depression; Anxiety
Keywords: Mindfulness; MBI; Depression; Anxiety disorders; Virtual; Short-term
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The experimental design is a RCT with two conditions: 1) treatment condition and 2) wait-list control condition. Outcome measures will focus on self-reported ratings of (primary) depression, anxiety, and stress and (secondary) well-being measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-based intervention (Experimental): Participants will take part in an adapted and abbreviated version of the traditional eight-week MBCT protocol, conducted virtually via Zoom. Participants will meet for five, weekly, two-hour sessions. The group size will be larger than traditional MBCT groups (i.e. 16-20 participants rather than 12 participants).
  Interventions: Behavioral: Mindfulness-Based Intervention
- Waitlist (No Intervention): Participants will be placed in a group with no treatment interventions for the duration of five weeks. Once these five weeks are complete, these participants will be placed in the next mindfulness clinic session to receive treatment. This does not the typical wait-list time for clinical services, which currently exceeds eight weeks

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — Mindfulness practices use a non-stigmatizing approach, combining secularized eastern meditative practices with western psychological advances to improve stress-management and self-care. Participants learn to generate less distress, engage more positively and fully in their lives and experiences, and respond more adaptively to challenges instead of reacting in automatic and unhelpful ways.
  Arms: Mindfulness-based intervention

SUMMARY:
Mindfulness-based interventions (MBIs) have emerged as clinically effective interventions for anxiety, depression, and general distress. However, there are significant barriers to accessing MBIs in the general population including length of treatment and cost. Furthermore, in the present COVID-19 pandemic, there is a demand to conduct virtual clinical services. However, to date, not much is known regarding the effectiveness of mindfulness groups that are conducted virtually. The aim of the present study is to examine the effectiveness of a five-week abbreviated MBCT intervention delivered virtually for a physician-referred, treatment-seeking, community sample. The virtual mindfulness group will be compared to a five-week wait-list control group. All wait-listed study participants will be given the opportunity to participate in the intervention after study completion. At present, clinical wait times for services far exceed five weeks, thus participants that are wait-listed will not experience delay in their treatment.

DETAILED DESCRIPTION:
Symptoms of depression and anxiety are extremely prevalent in the population. Unfortunately, patients often face barriers to accessing mental health care, particularly psychotherapeutic interventions, including long wait-times and demanding therapeutic protocols. For instance, standardized MBIs such as mindfulness-based cognitive therapy (MBCT) and mindfulness-based stress reduction (MBSR) are typically eight weeks in length. MBSR and MBCT, traditional MBTs, can demand over 30 hours of clinical time, and 50-60 hours of homework, all of which can be barriers to care. Furthermore, many clients are unable to access in-person interventions. At present the Sunnybrook Mindfulness Clinic is not conducting any virtual services due to the unknown benefit of virtual mindfulness interventions, creating significant barriers to clinical care for patients. The goal of this project is to compare the effectiveness of virtually delivered, abbreviated MBI (<10 hours of clinical time and <10 hours of homework) to a wait-list control condition in terms of reducing symptoms of depression/anxiety/stress and improving wellbeing. If effective, this abbreviated MBI conducted virtually could enable clients to pursue virtual services during the current COVID-19 pandemic.

MBTs use a non-stigmatizing approach, combining secularized eastern meditative practices with western psychological advances to improve stress-management and self-care. Participants learn to generate less distress, engage more positively and fully in their lives and experiences, and respond more adaptively to challenges instead of reacting in automatic and unhelpful ways. Participants in MBI often describe the intervention as transformative. The abbreviated MBI protocol has been piloted in an uncontrolled study and indicated significant benefit for patients in terms of symptom improvement. However, this will be the first time that the investigators pilot a virtual adaptation to the mindfulness group.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* are referred to the mindfulness group by a physician

Exclusion Criteria:

* have previously completed a full (≥8-week) MBI in the past 3 years
* meet criteria for substance abuse, psychosis, and/or mania
* express active suicidality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder - 7 (GAD-7) | At Baseline (week 0), Mid-treatment (week 3) and post-treatment (week 5) over five week intervention period.
  The GAD-7 is a 7-item self-report measure that assesses the presence of generalized anxiety symptoms within previous two weeks. Measure will be used to assess change in presence of generalized anxiety symptoms at baseline, mid-treatment, and post-treatment. Response options for the 7-item scale range from 0 (Not at All) to 3 (Nearly every day), and scale scores range can from 0 to 21.
Depression, Anxiety, Stress Scale-21 (DASS-21) | At Baseline (week 0), Mid-treatment (week 3) and post-treatment (week 5) over five week intervention period.
  The DASS-21 is a 21-item measure used to assess depression, anxiety, and stress symptoms. Measure will be used to assess change in presence of depression, stress, and anxiety symptoms at baseline, mid-treatment, and post-treatment. The DASS-21 is a shortened version of the original DASS, which was 42 items in length.
Patient Health Questionnaire - 9 (PHQ-9) | At Baseline (week 0), Mid-treatment (week 3) and post-treatment (week 5) over five week intervention period.
  The PHQ-9 is a 9-item measure for assessing depression severity. Measure will be used to assess change in depressive severity at baseline, mid-treatment, and post treatment.
  PHQ-9 scores can range from 0 to 27, as each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day)

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | At three time points (weeks 0,3, and 5) over 5 week intervention period.
  The Perceived Stress Scale (PSS) is a 10-item measure that assesses perceived stress within the last month. It is frequently used as a measure of acute distress, thus this measure is expected to be inversely related to positive well-being.
Warwick Edinburgh Mental Well- Being Scale (WEMWBS) | At three time points (weeks 0,3, and 5) over 5 week intervention period.
  The Warwick Edinburgh Mental Well- Being Scale (WEMWBS) is a 14-item measure that assesses positive well-being within the last two weeks.
Self-Compassion Scale | At three time points (weeks 0,3, and 5) over 5 week intervention period.
  The Self-Compassion Scale is a 24-item scale that assesses an individual's level of self-compassion.
Five Facet Mindfulness Questionnaire (FFMQ) | At three time points (weeks 0,3, and 5) over 5 week intervention period.
  The FFMQ is a 39-item questionnaire that assesses an individual's self-perceived use of mindfulness in their daily life.
Maslach Burnout Inventory (MBI) | At three time points (weeks 0,3, and 5) over 5 week intervention period.
  The MBI is a 22-item questionnaire that assesses the frequency and intensity of perceived burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Rector, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No